CLINICAL TRIAL: NCT06256835
Title: A Randomized Controlled Study to Explore Effect of Myofascial Release on Dysphagia in Parkinson's Patients
Brief Title: Effect of Myofascial Release on Dysphagia in Parkinson's Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, PI, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Jinmo-Parkinson
Record Dates: First submitted 2024-02-03; First posted 2024-02-13 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Rehabilitation; Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental): Study lasts 21 days for each patient. All patients are given rehabilitation treatment.The experimental group was given the Myofascial Release Therapy, five days a week, once a day, for 30-60 minutes each time.
  Interventions: Behavioral: Rehabilitation treatment; Behavioral: Myofascial Release Therapy
- The control group (Active Comparator): Study lasts 21 days for each patient. All patients are given rehabilitation treatment, five days a week, once a day, for 30-60 minutes each time.
  Interventions: Behavioral: Rehabilitation treatment

INTERVENTIONS:
Behavioral: Rehabilitation treatment — Both groups are given rehabilitation treatment. The main intervention measures included: 1) non-invasive ventilator treatment, generally at least once every night and typically not exceeding continuous daily usage.; 2) attention to feeding and sleeping positions, with a recommended sleeping position of lateral recumbent and the head of the bed raised by 20-30°; 3) swallowing function training, such as tongue muscle stretching training, assisted anterior jaw protrusion training, lemon ice stimulation to the soft palate, pharyngeal wall, etc., generally 5 days per week, twice per day, 5-20 minutes each time; 4) pulmonary ultrashort wave therapy, generally at least 2-3 times a week, and not more than once a day; 5) physical therapy, such as intensive training for gross motor functions including lifting the head, turning over, sitting, crawling, standing, etc., generally 3-5 days per week, 1-2 times per day, 5-20 min each time.
Behavioral: Myofascial Release Therapy — Myofascial release, also known as fascial release or fascial manipulation, is a physical therapy used to treat muscle and fascial tissue tension or pain. It involves applying appropriate pressure and stretching to release tight fascia and soft tissues, improving blood circulation, alleviating pain, and promoting rehabilitation. Myofascial release therapy is commonly used to treat muscle spasms, chronic pain, skeletal and joint issues, among others.
  Arms: The experimental group

SUMMARY:
The goal of this clinical trial is to explore Clinical Effect of Myofascial Release Therapy in Dysphagic Parkinson's Patients. The main question it aims to answer is:

• Can Myofascial Release Therapy improve swallowing function in Parkinson's Patients? Patients will be randomly allocated into the control group or the experimental group, all under rehabilitation treatment, the experimental group will be given Myofascial Release Therapy. The study lasts 21 days for each patient. Researchers will compare the Functional Oral Intake Scale, Penetration-Aspiration Scale, Swallowing Quality of Life to see if the Myofascial Release Therapy can help improve the situation.

DETAILED DESCRIPTION:
Myofascial release, also known as fascial release or fascial manipulation, is a physical therapy used to treat muscle and fascial tissue tension or pain. It involves applying appropriate pressure and stretching to release tight fascia and soft tissues, improving blood circulation, alleviating pain, and promoting rehabilitation.

The goal of this clinical trial is to explore Clinical Effect of Myofascial Release Therapy in Dysphagic Parkinson's Patients. The main question it aims to answer is:

• Can Myofascial Release Therapy improve swallowing function in Parkinson's Patients? Patients will be randomly allocated into the control group or the experimental group, all under rehabilitation treatment, the experimental group will be given Myofascial Release Therapy. The study lasts 21 days for each patient. Researchers will compare the Functional Oral Intake Scale, Penetration-Aspiration Scale, Swallowing Quality of Life to see if the Myofascial Release Therapy can help improve the situation.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Meeting the diagnostic criteria for Parkinson's disease.
* Diagnosed with dysphagia confirmed by the video fluoroscopic swallowing study.
* Water swallow test> Level 3.
* Stable vital signs, conscious, able to cooperate with assessment and treatment.

Exclusion Criteria:

* Dysphagia possibly caused by other reasons, such as cerebrovascular disease, trauma, neuromuscular diseases, malignant diseases of the pharynx and larynx, and digestive tract diseases.
* Complicated with cognitive impairment or consciousness dysfunction.
* Simultaneously suffering from severe liver, kidney failure, tumors, or hematological diseases.
* Complicated with severe liver and kidney failure, tumors, or hematological disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale | day 1 and day 21
  Penetration-Aspiration Scale was used to assess dysphagia under Videofluoroscopic Swallowing Study, primarily evaluating the extent to which fluid food entered the airway and caused penetration or aspiration during the swallowing process. The scores ranged 1 point to 8 points. As the level increased, the severity of dysphagia also increased.

SECONDARY OUTCOMES:
Swallowing Quality of Life questionnaire | day 1 and day 21
  Swallowing Quality of Life questionnaire was used to evaluate the quality of life, which consists of 44 items and divided into 11 main domains, including: overall satisfaction, understanding, diet, hydration, communication, respiratory issues, postoperative recovery, social impact, mental health, saliva control, and appearance. The maximum rough score was 220 points, which was converted into a standard percentage system in our study. As the scores increased, the quality of life was better.
patient health questionnaire-9 | day 1 and day 21
  The depression of the patients was evaluated with the patient health questionnaire-9. The scores ranged 0-27. As the scores increased, the severity of depression also increased.
Functional Oral Intake Scale | day 1 and day 21
  During Dysphagia-Functional Oral Intake Scale assessment, evaluators engage in communication with the patient, conduct observations, and make records to assess the patient's oral intake ability. The Functional Oral Intake Scale assessment form includes seven levels of scoring, ranging from level 1 to level 7, indicating a progressive improvement in the patient's oral intake ability. In general, the result below level 6 indicates unsafe for oral intake while level 6 and above indicates that eating via mouth can be safely conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Principal Investigator — Site Coordinator of United Medical Group located in Miami

IPD SHARING:
Plan to Share IPD: No